CLINICAL TRIAL: NCT05325983
Title: Using Saliva Stimulation to Immediately Improve Heart Failure Inpatient's Thirst Sensation: A Double-blind, Randomized Control Trial
Brief Title: Using Saliva Stimulation to Immediately Improve Heart Failure Inpatient's Thirst Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LI-JU Chen (Other)
Responsible Party: Sponsor-Investigator, LI-JU Chen, Investigator, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201901556B0
Record Dates: First submitted 2022-01-25; First posted 2022-04-13 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure; Thirst; Saliva
Keywords: Heart Failure; Thirst; Saliva stimulation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lemonade ice cubes (Experimental): 10 ml lemonade ice cubes in mouth, 45 seconds, 90 seconds, 135 seconds, 180 seconds respectively
  Interventions: Other: lemonade ice cubes
- water ice cubes (Placebo Comparator): 10 ml water ice cubes in mouth, 45 seconds, 90 seconds, 135 seconds, 180 seconds respectively
  Interventions: Other: water ice cubes

INTERVENTIONS:
Other: lemonade ice cubes — Mixing 1 part lemon juice and 6 parts boiling water, make 10ml lemonade ice cubes. The experimental group was given a 10ml lemonade ice cube. The ice cubes were weighed first and then given. The subjects were required to hold the lemonade ice cube in their mouths without breaking them, and not to swallow saliva. 45 seconds after the intervention is given, the nurse will use tweezers to take out the ice cube from the subject's mouth and weigh it , and then place the dry cotton swab at the opening of the sublingual gland in the oral cavity, take it out after 1 minute, and collect saliva, the recorded saliva volume = the collected saliva volume minus (10 ml ice cube weight minus the remaining ice cube weight); The experimental group was given a brand new 10ml lemonade ice cube. At 90 seconds, 135 seconds and 180 seconds, the above saliva collection method was repeated for a total of 5 times of saliva collection.
  Arms: lemonade ice cubes
Other: water ice cubes — make 10ml water ice cubes. The control group was given a 10ml water ice cube. The ice cubes were weighed first and then given. The subjects were required to hold the water ice cube in their mouths without breaking them, and not to swallow saliva. 45 seconds after the intervention is given, the nurse will use tweezers to take out the ice cube from the subject's mouth and weigh it , and then place the dry cotton swab at the opening of the sublingual gland in the oral cavity, take it out after 1 minute, and collect saliva, the recorded saliva volume = the collected saliva volume minus (10 ml ice cube weight minus the remaining ice cube weight); The control group was given a brand new 10ml water ice cube. At 90 seconds, 135 seconds and 180 seconds, the above saliva collection method was repeated for a total of 5 times of saliva collection.
  Arms: water ice cubes

SUMMARY:
The purpose of this study is to Using saliva stimulation to immediately improve heart failure inpatient's thirst sensation.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will screening period to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomize in a double-blind manner (participant and researcher) in a 1:1 ratio to experimental group (lemonade ice cubes) or the control group (water ice cubes).

ELIGIBILITY:
Inclusion Criteria:

* 1. Hospital stay for more than 24 hours;
* 2. NYHA III-IV;
* 3. Oral mucosa is intact, without ulcers or wounds;
* 4. Consciousness and normal cognitive function;
* 5. Those who are more than 20 years old and can answer the questionnaire in Chinese or Taiwanese verbally or in writing;
* 6. Normal swallowing function;
* 7. Stable vital signs and maintain systolic blood pressure above 90mmHg;
* 8. Those who need to limit water according to doctor's advice

Exclusion Criteria:

* 1. Those with endotracheal tube and respirator;
* 2. Those with indwelling nasogastric tube;
* 3. Those who fasted according to the doctor's advice;
* 4. Those who were diagnosed with dry syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Thirst intensity measured using an Visual Analogue Scale (VAS) | baseline and 180 second
  The VAS is a 100 mm line with anchor statements on the left (score :0 mm , no thirst) and on the right (score: 100 mm, extreme thirst).
  Change= (180 second score - baseline score)
Thirst distress measured using a Thirst Distress Scale-Heart Failure Taiwan version(TDS-HF) | baseline and 180 second
  The TDS-HF consists of 8 statements about how the patient experiences his/her thirst during the last 2-3 days (a total of 8 items). The 8 items are rated on a 5-point Likert scale. Patients are instructed to read each statement carefully and choose one of 5 possible answers for each statement that best describes the patients experience of thirst between strongly disagree (on the left side, number 1) and strongly agree (on the right side, number 5).
  Change= (180 second score - baseline score)
Change from Baseline in Measure Saliva Amount at 45 seconds. | baseline and 45 second
  Uses a dry cotton stick to place the sublingual gland opening in the subject's oral cavity for 1 minute, and collects the amount of saliva (baseline measurement; T0); then the intervention is performed Measures, 45 seconds (T1) after the intervention During the test, the nurse took out the ice cubes from the subject's mouth with tweezers and weighed it, and then placed the dry cotton swab at the opening of the sublingual gland in the oral cavity, took it out after 1 minute, and collected saliva. Weigh it with an electronic scale with a minimum weight of 0.01 grams, and assume that 1 gram is equal to 1 milliliter.
  Change= (45 second score - baseline score)
Change from Baseline in Measure Saliva Amount at 90 seconds. | baseline and 90 second
  Uses a dry cotton stick to place the sublingual gland opening in the subject's oral cavity for 1 minute, and collects the amount of saliva (baseline measurement; T0); then the intervention is performed Measures, 90 seconds (T2) after the intervention During the test, the nurse took out the ice cubes from the subject's mouth with tweezers and weighed it, and then placed the dry cotton swab at the opening of the sublingual gland in the oral cavity, took it out after 1 minute, and collected saliva. Weigh it with an electronic scale with a minimum weight of 0.01 grams, and assume that 1 gram is equal to 1 milliliter.
  Change= (90 second score - baseline score)
Change from Baseline in Measure Saliva Amount at 135 seconds. | baseline and 135 second
  Uses a dry cotton stick to place the sublingual gland opening in the subject's oral cavity for 1 minute, and collects the amount of saliva (baseline measurement; T0); then the intervention is performed Measures, 135 seconds (T3) after the intervention During the test, the nurse took out the ice cubes from the subject's mouth with tweezers and weighed it, and then placed the dry cotton swab at the opening of the sublingual gland in the oral cavity, took it out after 1 minute, and collected saliva. Weigh it with an electronic scale with a minimum weight of 0.01 grams, and assume that 1 gram is equal to 1 milliliter.
  Change= (135 second score - baseline score)
Change from Baseline in Measure Saliva Amount at 180 seconds. | baseline and 180 second
  Uses a dry cotton stick to place the sublingual gland opening in the subject's oral cavity for 1 minute, and collects the amount of saliva (baseline measurement; T0); then the intervention is performed Measures, 180 seconds (T4) after the intervention During the test, the nurse took out the ice cubes from the subject's mouth with tweezers and weighed it, and then placed the dry cotton swab at the opening of the sublingual gland in the oral cavity, took it out after 1 minute, and collected saliva. Weigh it with an electronic scale with a minimum weight of 0.01 grams, and assume that 1 gram is equal to 1 milliliter.
  Change= (180 second score - baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: LI-JU Chen, Study Chair — Self
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan, Taiwan

IPD SHARING:
Plan to Share IPD: No